CLINICAL TRIAL: NCT06284044
Title: Facilitating Safe Transition to Home for Preterm Infants - a Retrospective Observational Study Using a National Database
Brief Title: Facilitating Safe Transition to Home for Preterm Infants - a National Database Study
Status: Completed | Type: Observational
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: NIHR204885
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2024-03

CONDITIONS: Premature Birth
Keywords: Discharge; Neonatal Intensive Care
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Preterm infants (i.e. born before 37 completed weeks of pregnancy) often require additional care and are admitted to neonatal units. Readiness for discharge home typically requires a level of physiological maturity, such that an infant is: 1) able to breathe spontaneously without additional support; 2) able to maintain body temperature; 3) able to take all nutritional requirements orally; 4) weighs ≥1700 grams and is consistently gaining weight.

Staying in the hospital longer than necessary can be detrimental to infants, stressful for families, and costly to the NHS. Reducing the length of stay by just one day would be meaningful to parents and could save the UK National Health Service (NHS) almost £25million per year. Currently little is known about whether, how long and why preterm infants stay in hospital beyond the point at which they are physiologically ready for discharge.

This study will use data from babies' medical records from the whole of England and Wales to identify the age and postmenstrual age when preterm infants reach each of the physiological barriers to discharge and identify which physiological discharge barrier requires preterm infants to remain in hospital the longest. The study will quantify the difference between the time preterm infants become physiologically ready for discharge and actual discharge home and describe factors associated with extended stays.

DETAILED DESCRIPTION:
Infants born preterm (i.e., before 37 completed weeks of pregnancy) often require additional care and are admitted to neonatal units. Depending on needs, preterm infants have varying lengths of hospital stay; most go home between 37 and 40 weeks' post-menstrual age. Before a preterm infant can go home, there must be a readiness for safe discharge. "Discharge readiness" typically requires a level of physiological maturity such that the infant can:

1. Breathe without support: preterm babies often have breathing pauses (apnoea of prematurity); many require breathing support. With maturity, infants can breathe without support. Some may continue to need additional oxygen, and some go home on oxygen therapy.
2. Maintain body temperature: initially preterm infants are nursed in incubators. As the ability to generate and preserve heat matures, infants may move into heated cots initially and then finally into regular cots with normal clothing and blankets.
3. Feed adequately: preterm infants can take time to establish feeding. Initially potentially needing parenteral nutrition. Milk is slowly introduced via a gastric tube. As the ability to suck and swallow matures, infants learn to feed orally (on the breast or by bottle). To be discharged without additional support, infants need to be able to take milk requirements orally. Occasionally, where the service is available, infants can go home with partial nasogastric feeding.
4. Gain weight: Most infants are considered ready if they weigh at least 1700-1800g and are consistently gaining weight.

In addition, families must be prepared to care for the infant independently (including keeping the baby warm, feeding, bathing, safe travel, and giving medicines) and be emotionally ready and confident.

Infants achieve maturity at variable pace and may become mature in some aspects but not all e.g., be able to breathe well, maintain temperature, and gain weight, but still be unable to take sufficient oral feeds. The final reason that keeps the infant in hospital is referred to as the "terminal or final discharge barrier". There is very little research to investigate the barriers to safe discharge and to find the most common "final discharge barrier" for preterm infants in the UK.

The study team will use data from the National Neonatal Research Database (NNRD) for all infants born at <37 weeks' gestational age and admitted to neonatal units in England and Wales from 2016-2022. The day of life and postmenstrual age each infant reaches each of the physiological barriers to discharge will be described, and the final 'barrier to discharge' to be reached will be identified. The study team will assess whether the final discharge barriers differ by gestational age and between neonatal units and summarise the number of days infants remain in the hospital after surpassing all physiological milestones. The study team will explore the characteristics of infants, mothers and neonatal units that are associated with extended hospital stays beyond physiological readiness for discharge.

ELIGIBILITY:
Inclusion Criteria:

* Infants admitted to neonatal units that contribute data to the NNRD who are:
* Born at <37 completed weeks' gestational age
* Born from 01 January 2016 to 31 December 2022
* Admitted to neonatal care for >48 hours
* Discharged home alive

Ages: 22 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will include all infants born at <37 weeks gestational age who are admitted to a neonatal unit in England and Wales which contributes data to the National Neonatal Research Database (NNRD).
Sampling Method: Probability Sample
Enrollment: 250000 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Age and postmenstrual age when each of three physiological barriers are reached | 01 January 2016 to 31 December 2022
  Age (in days of life) and postmenstrual age (e.g., 35 weeks + 1 day) when each of three physiological barriers reached:
  1. Breathing spontaneously without having received caffeine (used to treat apnoea) for at least 5 days
  2. Achieved full oral feeding without need for intravenous or gastric feeding
  3. Weight ≥1700 grams
Final barrier to discharge home | 01 January 2016 to 31 December 2022
  The last of three physiological barriers to be surpassed

SECONDARY OUTCOMES:
Number of days in hospital after surpassing all physiological discharge barriers | 01 January 2016 to 31 December 2022
  Difference (in days) between reaching the last of the three physiological barriers to be reached and the day of discharge home

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Ojha, PhD, Study Chair — University of Nottingham
Locations (1):
- University Hospitals of Derby and Burton, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Szatkowski L, Abramson J, Tao S, Seaton SE, Dorling J, Arellano-Meza M, Harvey J, Harvey T, Ojha S. Facilitating safe transition to home for preterm infants (FAST home): Protocol for a retrospective observational study. PLoS One. 2025 Feb 11;20(2):e0318309. doi: 10.1371/journal.pone.0318309. eCollection 2025. PMID 39932978